CLINICAL TRIAL: NCT02455362
Title: A Multi-site, Double-blind, Parallel Arm, Block Randomised, Placebo Controlled, Factorial Phase III Study of Opioids for Chronic Refractory Breathlessness in People With Chronic Obstructive Pulmonary Disease.
Brief Title: Opioids for Refractory Breathlessness in Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: 'Recruitment not possible given changes to trial criteria
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, David Currow, Professor, Flinders University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 022/13 V.3.2.3
Record Dates: First submitted 2015-04-20; First posted 2015-05-27 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Placebo (Placebo Comparator): Double-blind placebo capsule, looking identical to capsules with active treatment, during all three treatment weeks.
  Interventions: Drug: Placebo
- Morphine sulfate (0, 0, 8 mg) (Experimental): Placebo during treatment week one and two and morphine 8 mg per day week three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (0, 8, 8 mg) (Experimental): Placebo during treatment week one and morphine 8 mg per day week two and three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (0, 8, 16 mg) (Experimental): Placebo week one, morphine 8 mg per day week two, and morphine 16 mg per day week three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (8, 8, 8 mg) (Experimental): Morphine 8 mg per day during all three treatment weeks.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (8, 8, 16 mg) (Experimental): Morphine 8 mg per day week one and two and morphine 16 mg per day week three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (8, 16, 16 mg) (Experimental): Morphine 8 mg per day week one and morphine 16 mg per day week two and three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (8, 16, 24 mg) (Experimental): Morphine 8 mg per day week one, morphine 16 mg per day week two, and morphine 24 mg per day week three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (16, 16, 16 mg) (Experimental): Morphine 16 mg per day during all three treatment weeks.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (16, 16, 24 mg) (Experimental): Morphine 16 mg per day week one and two, and morphine 24 mg per day week three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (16, 24, 24 mg) (Experimental): Morphine 16 mg per day week one and morphine 24 mg per day during week two and three.
  Interventions: Drug: Morphine sulfate
- Morphine sulfate (16, 24, 32 mg) (Experimental): Morphine 16 mg per day week one, morphine 24 mg per day week two, and morphine 32 mg per day week three.
  Interventions: Drug: Morphine sulfate

INTERVENTIONS:
Drug: Morphine sulfate — Treatment with sustained-release morphine sulfate is given as one double-blind capsule in the morning.
  Other Names: Kapanol(R)
  Arms: Morphine sulfate (0, 0, 8 mg); Morphine sulfate (0, 8, 16 mg); Morphine sulfate (0, 8, 8 mg); Morphine sulfate (16, 16, 16 mg); Morphine sulfate (16, 16, 24 mg); Morphine sulfate (16, 24, 24 mg); Morphine sulfate (16, 24, 32 mg); Morphine sulfate (8, 16, 16 mg); Morphine sulfate (8, 16, 24 mg); Morphine sulfate (8, 8, 16 mg); Morphine sulfate (8, 8, 8 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Breathlessness, the sensation of breathing discomfort, is a major problem in people with chronic obstructive pulmonary disease (COPD). Breathlessness that persists despite optimal management of the underlying disease(s) is said to be refractory.

Preliminary evidence suggests that a small, regular dose of morphine helps to reduce safely the sensation of breathlessness. However, this research on morphine for breathlessness has not defined the best way to adjust the dose of the medication, or refined which people are most likely to have benefit, no response or side effects.

This is a randomized, double-blind phase III trial in people with COPD and significant refractory breathlessness, which will explore several important questions:

* Are regular, low dose opioids (morphine) at four possible doses over 3 weeks more effective than placebo medication (containing no active ingredient) at improving breathlessness?
* Does the medication have any effect on daily activity, breathlessness, and quality of life?
* What are the common side effects of this intervention?
* Does the benefit from the drug outweigh the side effects it produces?
* Are there specific characteristics of people who are more likely to receive benefit from sustained release morphine?

Participants will be allocated to receive three weeks of morphine sulfate (and laxative, docusate with senna), or placebo (and placebo laxative). The dose of morphine may be increased each week for weeks two and three. All medicines will appear the same (blinded) and neither the doctor nor the participant will know which medication the participant is receiving.

Participants will have a medical interview, physical examination to collect some general health information, and baseline measurements including; daily activity, symptoms, and quality of life. A small amount of blood may be required to check eligibility. Further blood samples may be taken at week 1 and 3 to enable testing on how individuals respond to opioids, further consent will be obtained for these samples. Data on benefits, side effects, and medical care will be collected during comprehensive weekly visits. Participants will also fill out a simple diary twice daily for weeks one to three of the study, and for one day each week during an optional 3 month extension stage.

The outcome of this study may enable better management of symptoms and activity in people COPD with medicines that are shown to be effective and safe.

DETAILED DESCRIPTION:
Background: Three hundred thousand (300,000) Australians are breathless at rest or on minimal exertion, often for years, despite optimal treatment of the underlying cause(s). This includes more than 70,000 people who are too breathless to leave their homes often for long periods of time. Underlying causes for such severe and ongoing breathlessness include chronic obstructive pulmonary disease (COPD), interstitial lung disease, heart failure, neurodegenerative diseases such as motor neurone disease and cachexia from any cause. The prevalence of chronic refractory breathlessness will continue to increase as the population ages because the chronic progressive diseases where breathlessness is common are increasing in prevalence. Nearly one half of all people experience distressing breathlessness during the last year of life.

The American Thoracic Society defines breathlessness as "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity". The term 'dyspnoea' is used interchangeably with breathlessness, shortness of breath, breathing difficulty and laboured breathing.

Internationally, no medication is registered for the symptomatic reduction of chronic refractory breathlessness despite recommendations from the American Thoracic Society, the American College of Physicians, the Canadian Thoracic Society and the American College of Chest Physicians that regular, low-dose morphine is the evidence-based pharmaceutical option.

Aim: To enhance the evidence base for the pharmacological treatment of chronic refractory breathlessness using potential therapies compared to placebo.

Primary objective: To compare the difference of the net clinical effect (benefits and side effects) on chronic refractory breathlessness in people with chronic obstructive pulmonary disease (COPD) taking once daily, sustained release morphine at two different doses when compared to placebo.

Secondary objectives.

1. Are regular, low dose oral opioids safe, including when the dose is titrated upwards, in a population of people with refractory breathlessness and COPD?
2. Do people whose breathlessness is helped by regular, low dose oral morphine get additional benefit by further increasing the dose of morphine?
3. Over what period of time does benefit continue to increase once a dose level with benefit is achieved?
4. What percentage of people derive clinically significant benefit at each of four dosing levels over and above placebo?
5. At the lower doses, is there evidence that any benefit does not last the full 24 hours? (end-of-dose failure)
6. Can we predict response, benefit and side effects from baseline demographic and clinical data
7. Does the treatment of breathlessness with regular, low dose morphine have any effect on general health status and quality of life?
8. Determine if there is a change in activities of daily living in those treated with opioids when compared to placebo.
9. Assess any effects of each treatment on anxiety and depression.
10. Understand the longer term benefits and side effects from sustained release morphine in people with COPD when compared to placebo.
11. Do participants, while still blinded, have any preference at the end of the three week study?

Sub-studies

1. Identify pharmacokinetic and pharmacodynamic parameters that may help to predict which individuals will achieve the greatest benefit in week one of therapy (8mg/day, 16mg/day).
2. Identify pharmacogenomic variations in opioid receptors and signaling that may help to predict clinical response (benefit, side effects or no response).
3. Study the effect on sleep in people participating in the study
4. Compare the within trial incremental cost and cost effectiveness of the therapy
5. Evaluate any changes in total testosterone from baseline to the end of the three month extension.

Null hypothesis: In people who have COPD with refractory breathlessness, there is no difference in breathlessness intensity with the addition of regular, low dose oral sustained release morphine when compared to placebo.

Alternative hypothesis: The addition of regular, low dose oral sustained release morphine reduces the intensity of breathlessness in people with COPD and that this occurs safely.

Study design:

A five stage, national, multi-site, double-blind, parallel arm, block randomised, placebo controlled factorial (dose increment) phase III study of opioids for chronic refractory breathlessness in people with COPD:

Stage 0 - baseline (2 days); Stage 1 - randomisation #1 (1 week); Stage 2 - randomisation #2 (1 week); Stage 3 - randomisation #3 (1 week); and Stage 4 - an optional blinded extension arm (up to 3 months).

Stage 0. Baseline assessment: All consenting participants will complete 2 full days of baseline diary (morning and evening) in order to become accustomed to completing the diary regularly and to provide stable baseline data regarding breathlessness, symptoms and function (as measured by activPALR actigraphy). At completion of the 2 days, the participant will be reviewed, complete the remaining baseline assessments (questionnaires, measures and baseline safety data), and will then be eligible to be randomised the first time.

Time period: Two full days (4 diary entries)

Stage 1. Randomisation #1: Randomisation to mane orally: placebo OR 8mg KapanolR OR 16mg KapanolR. Twice daily diary. Participants randomised to KapanolR will also receive blinded docusate with sennosides, while those randomised to placebo will receive identical placebo. This is the primary outcome (end point) of the study.

Time period: 1 week

Stage 2. Randomisation #2: While continuing the arm assigned in Stage 1, add a randomisation to mane orally: placebo OR 8mg KapanolR. Twice daily diary. Participants who were randomised to placebo in Stage 1 and KapanolR in Stage 2 will have blinded docusate with sennosides replace placebo.

Time period: 1 week

Stage 3. Randomisation #3: While continuing the arm assigned in Stages 1 and 2, add a third randomisation to mane orally: placebo OR 8mg KapanolR. Twice daily diary. activPALR accelerometer worn this week. Participants who were randomised to placebo in Stages 1 and 2 and KapanolR in Stage 3 will have blinded docusate with sennosides replace placebo.

Time period: 1 week

Stage 4. Extension (optional for each individual participant): Continue double blind medications from Stages 1, 2 and 3 for up to three months. Diary one day each week. A blood test at the end of the three months will be taken for total testosterone levels.

Time period: up to 3 months.

Target population: This study is for people with optimally treated people with mild, moderate or severe chronic obstructive pulmonary disease (COPD).

Primary outcome and its assessment: Change from baseline average intensity of breathlessness over the previous 24 hours, measured each morning on a 11 point numerical rating scale.

Significance: The study will answer several practical questions including whether opioids have a net benefit in people with COPD in reducing refractory breathlessness, whether dose increases beyond initial response provide a greater net benefit, the pattern of symptomatic response in the days after successful titration, and the proportion of people who derive a clinically meaningful symptomatic benefit at each dose level.

Analysis plan: All analyses will be conducted on an intention-to-treat basis. All analyses will be conducted with Stata version 13.1. Missing data will be imputed using multiple imputation with 50 resamples drawn. The primary comparisons on which the study is powered are at the end of week 1: placebo compared to 8mg KapanolR daily; and placebo compared to 16mg KapanolR daily. Change in breathlessness in the first week between these groups will be evaluated using a random effects mixed model.

Sample size calculations: All calculations assume Type I (familywise error rate (FWER)) error rate of 5% and Type II error rate of 20% (power of 80%) respectively. In order to account for attrition of 20% by the end of week 1, the study will recruit 144*100/ (100-20) = 180 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Physician diagnosed COPD confirmed by spirometry, defined as a prior post-bronchodilator FEV1/FVC < 0.7 in accordance with the GOLD 2014 criteria
* On stable medications relating to the optimal treatment of COPD or its symptomatic management over the prior week except routine "as needed" medications.
* Breathlessness of a level two (2) or higher on the modified Medical Research Council (mMRC) dyspnoea scale
* English speaking with sufficient reading and writing ability to complete the study questionnaires
* Assessed as competent (using SLUMS score of 27 for high school, and 25 for less than high school)
* Able and willing to give written informed consent

Exclusion Criteria:

* On regularly prescribed opioid medications, including codeine preparations at or above 8mg oral morphine equivalent daily in the previous seven (7) days.
* History of adverse reactions to any of the study medications or constituents in the placebo;
* Australian-modified Karnofsky performance score (AKPS) less than 50 at the beginning of the study.
* Respiratory or cardiac event in the previous one week (excluding upper respiratory tract infections). Illness must have resolved completely prior to baseline evaluation, as judged by the person's treating physician.
* Evidence of respiratory depression with resting respiratory rate <8/min.
* Documented central hypoventilation syndrome.
* Chronic alcoholism, or previous or recent history of substance misuse.
* Uncontrolled nausea, vomiting or evidence of a gastrointestinal tract obstruction.
* Renal dysfunction with creatinine clearance calculated (MDRD) less than 20 mls/minute.
* Evidence of severe hepatic impairment defined as transaminases or bilirubin >4x normal (Excluding Gilbert's syndrome)
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline intensity of breathlessness over the previous 24 hours | Week 1
  Rated on a 0-10 numerical rating scale (NRS) in a diary each evening. The primary endpoint is the difference between placebo, morphine sulfate 8 mg, or 16 mg after the first treatment week.

SECONDARY OUTCOMES:
Change from baseline unpleasantness of breathlessness over the previous 24 hours | Week 3
  Rated on a 0-10 numerical rating scale (NRS) in a diary each evening.
Change from baseline intensity of breathlessness "right now" | Week 3
  Rated on a 0-10 numerical rating scale (NRS) in a diary each morning.
Change from baseline in the intensity of breathlessness | Week 1
  In addition to the NRS ratings, the intensity of breathlessness is rated on a 0-10 modified Borg scale in a evening diary.
Current medication use and compliance | At study end for up to 15 weeks.
  Collected in a diary in the evening, including of any rescue medication used.
Number of participants with adverse events | At study end for up to 15 weeks.
  Collected in a diary in the evening.
Change from baseline physical activity using an accelerometer | Week 3
  Measured during two days at baseline and during at least five days of treatment week three.
Change from baseline in concurrent symptoms | Week 1
  Measured using the revised Edmonton Symptoms Assessment Scale (ESAS-r).
The modified Medical Research Council (mMRC) breathlessness scale | At study end for up to 15 weeks.
  Measures the functional impact of breathlessness.
Change from baseline serum testosterone level | At the end of the 3 month follow-up stage, after up to 15 weeks.
  To explore whether longer term morphine treatment is associated with decreased levels of testosterone.
Change from baseline pharmacogenomic opioid blood profile | Week 1
  From the baseline sample, the UGT2B7*2 and *28 polymorphisms, P-glycoprotein (ABCB1 5SNPs in a haplotype block), the 5-hydroxytryptamine type 3B (HTR3B) gene rs7103572, and mu opioid receptor (A118G) polymorphisms will be measured. Interleukin 1ß, TNFalpha and Il-6 will be measured at baseline and at the end of the first treatment week.
Pharmacodynamic/-kinetic blood samples | Week 1
  In a subset of 55 participants, blood parameters for morphine and its metabolites will be analysed (4 blood samples over 8 hours) at steady state of the treatment at the end of the week 1.
Change from baseline end-tidal carbon dioxide | Week 3
  Exhaled gas measured using a non-invasive capnometer.
Change from baseline pulse oximetry | Week 3
  Non-invasive measurement of the oxygen saturation, respiratory rate, and heart rate.
Change from baseline sleep quality | The final night of week 3
  Twenty (20) participants at the Sydney and Adelaide sites will be invited to undertake a simple, non-invasive home sleep study using the ResMed ApneaLink Plus device.
Change from baseline sleep quality | During the study for up to 15 weeks.
  Rated on a 4 point Likert scale in a morning diary.
Change from baseline sleep quality and sleep-related problems | Week 3
  The questionnaires used are the Epworth Sleepiness Scale, Leeds Sleep Questionnaire, and the Karolinska Sleepiness Scale.
Change from baseline bowel function index | Week 1
  Measure of the bowel function, during treatment with placebo / morphine sulfate 8 or 16 mg.
Change from baseline breathlessness-related quality of life | Week 3
  Measured on the CRQ-SAS Dyspnoea sub-scale.
Change from baseline health-related quality of life | During the study for up to 15 weeks.
  Measured using the EQ-5D questionnaire.
Change from baseline Life-space | During the study for up to 15 weeks.
  Life-Space is a measure of where a person goes, the frequency of going there, and the dependency in getting there.
Change from baseline Australian Karnofsky Performance Status | During the study for up to 15 weeks.
  A score of 0 to 100 (in increments of 10) is assigned to participants based on their ability to undertake a range of daily tasks. The score gives an indication of the participant condition in terms of physical ability.
Change from baseline Hospital Anxiety and Depression Scale | Week 3
  A 14-item questionnaire used to measure anxiety and/or depression.
Global Impression of Change | During the study for up to 15 weeks.
  Participant-rated seven point scale of the perception of their change, specifically their improvement since the commencement of the study.
Blinded patient preference to continue treatment | At study end after up to 15 weeks.
  Participants will be asked for their preference to continue at study exit ('Is this a therapy which, on balance, you would continue to take for your breathlessness?')
Health economy composite | During the study for up to 15 weeks.
  Data on all health care contacts including lenght of hospitalizations, emergency department visits, DRG codes, outpatient visits to general practitioner and community nurse, and date of death.

CONTACTS AND LOCATIONS:
Overall Officials: David C Currow, MD, PhD, Principal Investigator — Flinders University